CLINICAL TRIAL: NCT01988012
Title: An Open-label, Multicenter Study to Evaluate Disease Activity and Safety of Treatment With Actemra (Tocilizumab) Administered as Subcutaneous Injection in Adult RA Patients.
Brief Title: A Study of the Efficacy and Safety of Tocilizumab in Adults With Rheumatoid Arthritis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28698
Record Dates: First submitted 2013-10-31; First posted 2013-11-20 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Adults with rheumatoid arthritis will be treated with tocilizumab for 24 weeks followed by an 8 week follow-up period without treatment.
  Interventions: Biological: tocilizumab

INTERVENTIONS:
Biological: tocilizumab — 162 milligram (mg) administered subcutaneously once weekly for 24 weeks
  Other Names: RoActemra/Actemra

SUMMARY:
A multi-center, open-label single-arm study to evaluate the efficacy and safety of tocilizumab administered as a single, weekly injection in adults with rheumatoid arthritis. Combination therapy with methotrexate or other non-biologic disease modifying anti-rheumatic drugs (DMARDs) was permitted.

ELIGIBILITY:
Inclusion Criteria:

* Adults >/= 18 years of age
* Diagnosis of active rheumatoid arthritis (RA) according to the revised (1987) American College of Rheumatology (ACR) criteria or European League Against Rheumatism (EULAR)/ACR (2010) criteria
* Previously treated with the following: three non-biologic DMARDs, and not treated with any biologic agent OR one biologic agent (alone or in combination with non-biologic DMARDs), and discontinued that agent for a reason
* Oral corticosteroids (</= 10 mg/day prednisone or equivalent), non-steroidal anti-inflammatory drug (NSAIDs) and non-biologic DMARDs are permitted if on a stable dose regimen for >/= 4 weeks prior to Baseline
* Use of effective contraception throughout the study as defined by protocol; female patients of childbearing potential must not be pregnant

Exclusion Criteria:

* Presence of serious, uncontrolled, clinically significant medical conditions
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower gastrointestinal (GI) disease that might predispose to perforation
* Current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections
* Any infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks of Screening or oral antibiotics within 2 weeks of Screening
* Clinically significant findings on lab tests and/or hepatitis B or C, or human immunodeficiency virus (HIV) screenings
* Active tuberculosis (TB) requiring treatments within the previous 3 years
* Evidence of active malignant disease, malignancies diagnosed within the previous 10 years, or breast cancer diagnosed within the previous 20 years
* History of alcohol, drug, or chemical abuse within 1 year prior to Screening
* Neuropathies or other conditions that might interfere with pain evaluation
* Major surgery (including joint surgery) within 8 weeks prior to Screening or planned major surgery within 6 months following Baseline
* Rheumatic autoimmune disease other than RA, including systemic lupus erythematosus, mixed connective tissue disorder, scleroderma, polymyositis, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's syndrome). Secondary Sjögren's syndrome with RA is permitted
* Functional Class IV as defined by the ACR Classification of Functional Status in-Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile RA, and/or RA before the age of 16
* Prior history of current inflammatory joint disease other than RA
* Exposure to tocilizumab (either IV or subcutaneous administration) at any time prior to Baseline
* Treatment with any investigational agent within 4 weeks (or five half-lives of the investigational drug, whichever is longer) of Screening
* Previous treatment with any cell-depleting therapies, including investigational agents approved therapies, with alkylating agents such as chlorambucil, or with total lymphoid irradiation
* Treatment with IV gamma globulin, plasmapheresis within 6 months of Baseline
* Immunization with a live/attenuated vaccine within 4 weeks prior to Baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Israel (8):
  - Beer Yaacov
  - Beersheba
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Adults with rheumatoid arthritis were treated with 162 milligram (mg) tocilizumab administered subcutaneously once weekly for 24 weeks. The protocol recommended suspending the treatment after week 24 for a period of 8 weeks, according to investigators' discretion, for the purpose of drug-free immunogenicity testing. In the present study, none of the participants had their tocilizumab treatment suspended.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 100
Completed | 85
Not Completed | 15
Not completed — Adverse Event | 5
Not completed — Insufficient Therapeutic Response | 3
Not completed — Patient Withdrawal of Consent | 4
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Groups:
- Tocilizumab: Adults with rheumatoid arthritis were treated with 162 mg tocilizumab administered subcutaneously once weekly for 24 weeks. The protocol recommended suspending the treatment after week 24 for a period of 8 weeks, according to investigators' discretion, for the purpose of drug-free immunogenicity testing. In the present study, none of the participants had their tocilizumab treatment suspended.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (11.8)
Gender [Count of Participants; unit: Participants]
  Female | 80
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Disease Activity Index (CDAI) Remission and CDAI Low Disease Activity
Description: Clinical Disease Activity Index (CDAI) is an index for measuring disease activity in rheumatoid arthritis (RA). The index was calculated using the following formula: CDAI = number of swollen joints using the 28-joint count (SJC28) + number of tender joints using the 28-joint count (TJC28) + patient global assessment of disease (PGA) based on 10 centimeter [cm] Visual Analog Scale [VAS] + physician global assessment of disease (PhGA) based on 10 cm VAS. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. Remission is defined as CDAI ≤2.8 and Low Disease Activity (LDA) is defined as 2.8< CDAI ≤10.
Time Frame: Week 24
Population: The analysis population included those participants from the full analysis set (FAS) for whom evaluable data for this outcome measure were available. The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 85
percentage of participants
  CDAI Remission | 16.5
  CDAI LDA | 34.1

2. Primary Outcome: Change From Baseline in CDAI
Description: Clinical Disease Activity Index (CDAI) is an index for measuring disease activity in rheumatoid arthritis (RA). The index was calculated using the following formula: CDAI = number of swollen joints using the 28-joint count (SJC28) + number of tender joints using the 28-joint count (TJC28) + patient global assessment of disease (PGA) based on 10 centimeter [cm] Visual Analog Scale [VAS] + physician global assessment of disease (PhGA) based on 10 cm VAS. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total CDAI scores ranged from 0 to 76, with higher scores indicating increased disease activity. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab. Here n is the number of participants with evaluable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  Baseline | 31.89 (14.35)
  Change from Baseline at Week 24: number analyzed (Participants) | 85
  Change from Baseline at Week 24 | -18.29 (14.52)

3. Primary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Remission and SDAI Low Disease Activity
Description: Simplified Disease Activity Index (SDAI) was an index for measuring disease activity in RA and had a good correlation with the DAS28. The index was calculated using the following formula: SDAI: SJC28 + TJC28 + PGA (10 cm VAS) + PhGA (10 cm VAS + C-Reactive Protein (CRP) in milligram/liter (mg/L). VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Scores ranged from 0 to 86, with higher scores also indicating increased disease activity. An SDAI score of ≤ 3.3 represents clinical remission, a score of ≤ 11.0 represents low disease activity.
Time Frame: Week 24
Population: The analysis population included those participants from the FAS for whom evaluable data for this outcome measure were available. The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 52
percentage of participants
  SDAI Remission | 19.2
  SDAI LDA | 38.5

4. Primary Outcome: Change From Baseline in SDAI
Description: Simplified Disease Activity Index (SDAI) was an index for measuring disease activity in RA and had a good correlation with the DAS28. The index was calculated using the following formula: SDAI: SJC28 + TJC28 + PGA (10 cm VAS) + PhGA (10 cm VAS + C-Reactive Protein (CRP) in mg/L. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Scores ranged from 0 to 86, with higher scores also indicating increased disease activity. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 98
units on a scale
  Baseline | 33.73 (14.83)
  Change from Baseline at Week 24: number analyzed (Participants) | 52
  Change from Baseline at Week 24 | -21.41 (14.99)

5. Primary Outcome: Change From Baseline in Disease Activity Score 28-Erythrocyte-Sedimentation Rate (DAS28-ESR)
Description: The DAS28-ESR score is a measure of the patient's disease activity calculated using the tender joint count on 28 joints (TJC28), swollen joint count on 28 joints (SJC28), patient's global assessment (PGA) of disease activity based on visual analog scale (VAS) and the erythrocyte sedimentation rate (ESR) in millimeter/hour (mm/hr). VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity). Total possible score ranged from 0 to 10. Higher scores represent higher disease activity. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 99
units on a scale
  Baseline | 4.98 (0.98)
  Change from Baseline at Week 24: number analyzed (Participants) | 84
  Change from Baseline at Week 24 | -2.47 (1.29)

6. Primary Outcome: Percentage of Participants Achieving 20%, 50% and 70% Improvement in American College of Rheumatology (ACR) Response Scores (ACR20, ACR50 and ACR70)
Description: An ACR20 response requires at least 20% improvement compared to baseline in SJC (based on 66 joints) and TJC (based on 68 joints) as well as at least 20% improvement in 3 of the following 5 assessments: 1) PGA pain VAS, 2) PGA VAS; 3) physician's global assessment of disease activity VAS, 4) Health Assessment Questionnaire-Disability Index (HAQ-DI) with 20 questions consisting of 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities, 0=without difficulty to 3=unable to do; and 5) CRP in mg/L or ESR in mm/hr. ACR50 and ACR70 responses are defined in a similar way except that they required a 50% and 70% improvement from baseline, respectively. VAS assessments involved a 10 cm horizontal scale from 0 (no disease activity) to 10 (maximum disease activity).
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 85
percentage of participants
  ACR20 | 62.4
  ACR50 | 37.6
  ACR70 | 20.0

7. Primary Outcome: Percentage of Participants With Good to Moderate European League Against Rheumatism (EULAR) Response
Description: Response was determined using EULAR criteria based upon DAS28 absolute scores at the assessment visit and the DAS28 reduction from the reference visit. Participants with a score lesser than or equal to (</=) 3.2 and reduction of greater than (>) 1.2 points were assessed as having a 'good' response. Participants with a score >3.2 with reduction of >1.2 points, or a score <=5.1 with reduction of >0.6 to <=1.2 points, were assessed as having a 'moderate' response. Participants with a score >5.1 with reduction of >0.6 to <=1.2 points, or any score with reduction <=0.6 points, were assessed as non-responders with response recorded as 'none.'
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 83
percentage of participants | 96.4

8. Primary Outcome: Change From Baseline in TJC and SJC
Description: The number of tender joints (based on 68 joints) and swollen joints (based on 66 joints) were counted at each visit. TJC was determined by identifying the joints that were painful under pressure or to passive motion; no tenderness =0, tenderness =1. SJC was determined by identifying swelling; no swelling =0, swelling =1. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
joint count
  TJC at Baseline | 21.42 (15.20)
  TJC Change from Baseline at Week 24: number analyzed (Participants) | 85
  TJC Change from Baseline at Week 24 | -11.91 (13.59)
  SJC at Baseline | 10.30 (10.27)
  SJC Change from Baseline at Week 24: number analyzed (Participants) | 85
  SJC Change from Baseline at Week 24 | -7.54 (9.60)

9. Primary Outcome: Change From Baseline in Percentage of Participants on Tocilizumab Monotherapy
Description: Participants were either on tocilizumab monotherapy or tocilizumab plus non-biologic disease modifying anti-rheumatic drugs (DMARDs). Reported here is the percentage of participants on tocilizumab monotherapy at baseline and the change from baseline at Week 24. A positive change from baseline at Week 24 indicates the percentage of participants, who discontinued DMARDs during the study.
Time Frame: Baseline, Week 24
Population: The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
percentage of participants
  Baseline | 26
  Change from Baseline at Week 24 | 12

10. Primary Outcome: Change From Baseline in Patient Global Assessment of Disease Activity Visual Analog Scale (PGA VAS)
Description: PGA VAS represents the participant's overall assessment of their current disease activity on a 100 millimeter (mm) horizontal VAS scale from 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  Baseline | 69.73 (24.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 85
  Change from Baseline at Week 24 | -31.22 (28.43)

11. Primary Outcome: Change From Baseline in Patient Pain VAS
Description: Patient Pain VAS represents the participant's assessment of his/her current level of pain on a 100 mm horizontal VAS scale from 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  Baseline | 64.82 (26.39)
  Change from Baseline at Week 24: number analyzed (Participants) | 85
  Change from Baseline at Week 24 | -29.11 (29.16)

12. Primary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI evaluates participant-reported quality of life using 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and other common activities and 20 questions. Each category contains multiple questions, which were answered using a 4-point scale from 0 (without any difficulty) to 3 (unable to do). The overall index score was an average of the individual item responses and may range from 0 to 3, where higher scores indicate more difficulty in daily living activities. A negative change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  Baseline | 1.55 (0.80)
  Change from Baseline at Week 24: number analyzed (Participants) | 85
  Change from Baseline at Week 24 | -0.34 (0.62)

13. Primary Outcome: Change From Baseline in Patient Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: The symptom-specific measure FACIT-F assesses chronic illness therapy with special emphasis on fatigue in the past 7 days and consists of 5 dimensions: 1) physical well- being, 2) social/family well-being, 3) emotional well-being, 4) functional well-being, and 5) additional concerns. Each of the questions is categorically answered using the scales 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much for a total possible FACIT-F score of 0 to 52. The figures are reversed during score calculations, so that higher score values indicate more favorable conditions. A positive change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  Baseline | 23.46 (11.32)
  Change from Baseline at Week 24: number analyzed (Participants) | 85
  Change from Baseline at Week 24 | 6.95 (9.70)

14. Primary Outcome: Total Scores on Hamilton Depression Rating Scale (HDRS) and Hamilton Anxiety Scale (HAS)
Description: The HDRS is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome. HAS is a clinician-administered assessment to measure the severity of anxiety symptoms and consists of 14 items with a total score range from 0 to 56. A higher score indicates a worse outcome.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
units on a scale
  HDRS at Baseline: number analyzed (Participants) | 77
  HDRS at Baseline | 7.87 (7.19)
  HDRS at Week 24: number analyzed (Participants) | 84
  HDRS at Week 24 | 4.94 (5.85)
  HAS at Baseline: number analyzed (Participants) | 77
  HAS at Baseline | 8.56 (8.43)
  HAS at Week 24: number analyzed (Participants) | 84
  HAS at Week 24 | 5.93 (7.17)

15. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and AEs of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant administered a drug and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug, whether or not considered related to the drug. Preexisting conditions which worsen during a study are also considered as AEs. AESIs are AEs that occur in categories of special interest with regard to the benefit-risk profile and overall safety of a drug. The following nine categories of AESIs were identified for tocilizumab: 1) serious and/or medically significant infections, 2) myocardial infarction/acute coronary syndrome, 3) gastrointestinal perforations, 4) malignancies, 5) anaphylaxis/hypersensitivity reactions, 6) demyelinating disorders, 7) stroke, 8) serious and/or medically significant bleeding events, and 9) serious and/or medically significant hepatic events.
Time Frame: Up to Follow-up Week 32
Population: The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
percentage of participants
  AEs | 70.0
  AESIs | 7.0

16. Secondary Outcome: Percentage of Participants Who Required Dose Modifications or Discontinued Study Due to AEs
Time Frame: Up to Week 24
Population: The FAS included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 100
percentage of participants
  % of Particpants with Dose Modifications | 16
  % of Participants Who Discontinued Study | 5

17. Secondary Outcome: Immunogenicity: Percentage of Participants With Anti-tocilizumab Antibodies
Description: Reported is the percentage of participants positive for anti-tocilizumab antibodies in the confirmatory anti-tocilizumab antibody assay, which followed an initial anti-tocilizumab screen. Participants, who withdrew from the study
Time Frame: Baseline, Week 24, Follow-up Week 32 and Early Withdrawal
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 97
percentage of participants
  Baseline | 1.0
  Week 24: number analyzed (Participants) | 85
  Week 24 | 0
  Follow-up Visit Week 32: number analyzed (Participants) | 76
  Follow-up Visit Week 32 | 0
  Early Withdrawal: number analyzed (Participants) | 10
  Early Withdrawal | 0

18. Secondary Outcome: Immunogenicity: Tocilizumab Levels
Time Frame: Week 12, Week 24, Follow-up Week 32 and Early Withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 91
microgram/milliliter (mcg/mL)
  Week 12 | 35.49 (17.81)
  Week 24: number analyzed (Participants) | 84
  Week 24 | 41.63 (22.79)
  Follow-up Week 32: number analyzed (Participants) | 59
  Follow-up Week 32 | 39.53 (28.47)
  Early withdrawal: number analyzed (Participants) | 9
  Early withdrawal | 19.04 (15.69)

19. Secondary Outcome: Immunogenicity: Change From Week 1 in Soluble Interleukin-6 Receptor (sIL-6R) Levels
Description: A positive change from Week 1 indicates an increase in sIL-6R levels.
Time Frame: Week 1, Week 12, Week 24, Follow-up Week 32 and Early Withdrawal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms/milliliter (ng/mL)
Arm/Group | Tocilizumab
Number analyzed (Participants) | 98
nanograms/milliliter (ng/mL)
  Week 1 | 38.33 (10.30)
  Change from Week 1 at Week 12: number analyzed (Participants) | 89
  Change from Week 1 at Week 12 | 475.79 (120.98)
  Change from Week 1 at Week 24: number analyzed (Participants) | 83
  Change from Week 1 at Week 24 | 503.67 (127.13)
  Change from Week 1 at Follow-up at Week 32: number analyzed (Participants) | 74
  Change from Week 1 at Follow-up at Week 32 | 382.26 (240.95)
  Change from Week 1 at Early withdrawal: number analyzed (Participants) | 10
  Change from Week 1 at Early withdrawal | 309.91 (183.07)

ADVERSE EVENTS:
Time Frame: Up to Follow-up Week 32
Description: The safety population included all enrolled participants who received at least one dose of subcutaneous tocilizumab.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 6/100
Other Adverse Events (participants affected / at risk) | 44/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=100)
Colitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Adnexal torsion (Reproductive system and breast disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=100)
Leukopenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 7
Alanine aminotransferase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 6
Hepatic enzyme increased (Investigations) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.